CLINICAL TRIAL: NCT00989001
Title: A Phase 3b Randomized, Double-Blind, Placebo Controlled, Parallel Group Study to Evaluate the Safety and Efficacy of Vernakalant Hydrochloride Injection in Patients With Recent Onset Symptomatic Atrial Fibrillation
Brief Title: A Phase 3b Study of Vernakalant Injection in Patients With Recent Onset Symptomatic Atrial Fibrillation (AF)(MK-6621-045)
Acronym: ACT V
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Advanz Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 6621-045; 6517-CL-0020 (Other: Merck); MK-6621-045
Record Dates: First submitted 2009-10-01; First posted 2009-10-02 (Estimated); Last update posted 2014-03-10 (Estimated); Status verified 2014-02

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation; RSD1235; Vernakalant; conversion
MeSH Terms: conditions — Atrial Fibrillation | interventions — vernakalant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vernakalant (Experimental): Maximum volume of 100 mL as per the dosing schedule, administered intravenously (IV) over 10 minutes
  Interventions: Drug: Vernakalant
- Placebo (Placebo Comparator): Placebo (saline) administered IV at same volume and rate as per dosing schedule for vernakalant
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vernakalant — Maximum volume of 100 mL as per the dosing schedule, administered intravenously (IV) over 10 minutes
  Other Names: RSD1235
  Arms: Vernakalant
Drug: Placebo — Injection
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of vernakalant injection in subjects with recent onset (AF > 3 hours to <= 7 days), symptomatic atrial fibrillation and no evidence or history of congestive heart failure.

DETAILED DESCRIPTION:
Participants received a 10-minute intravenous (IV) infusion of vernakalant (3 mg/kg) or an equivalent amount of normal saline (placebo), followed by a 15-minute observation period. If the participant was still in atrial fibrillation or atrial flutter, a second 10-minute IV infusion of vernakalant (2 mg/kg) or an equivalent amount of placebo was administered unless the participant experienced any dose-stopping criteria after the start of the first infusion. If a participant converted to sinus rhythm during the first or second infusion, that infusion was completed.

ELIGIBILITY:
Inclusion Criteria:

* Females must be not pregnant or nursing and if pre-menopausal, must be using an effective form of birth control from time of screening until 30 days post study treatment
* Subject must have recent onset (> 3 hours to <= 7 days) symptomatic AF to be best managed by acute conversion to SR
* Subject must have adequate anticoagulant therapy
* Subject must have systolic blood pressure (SBP) above 90 mmHg and less than 160 mmHg and diastolic blood pressure (DBP) less than 95 mmHg at screening and baseline
* Subject must have a body weight between 45 and 136 kg, inclusive (99 and 300 lbs)

Exclusion Criteria:

* Subject has a history of heart failure or documentation of left ventricular dysfunction
* Subject has known or suspected prolonged QT or uncorrected QT interval of > 0.440 sec
* Subject has symptomatic bradycardia or ventricular rate less than 50 bpm at Screening, unless controlled by a pacemaker
* Subject has bradycardia (heart rate less than 50 bpm) or hypotension (SBP less that 90 mmHg) after receiving a loading, bolus dose, or sustained infusion of any rate control medication during Screening
* Subject has a QRS interval > 0.14 sec., unless subject has a pacemaker
* Subject had a myocardial infarction (MI), acute coronary syndrome, cardiac surgery (including percutaneous transluminal coronary angioplasty (PTCA) or stent placement), within 30 days prior to enrollment or subject has evidence of new ischemic changes on Screening 12-lead ECG
* Subject has troponin I or T levels beyond the upper limit of normal for the local lab
* Subject has significant valvular stenosis, hypertrophic obstructive cardiomyopathy, restrictive cardiomyopathy or constrictive pericarditis
* Subject has failed electrical cardioversion for AF at anytime
* Subject has failed pharmacologic conversion with an intravenous Class I or Class III antiarrhythmic drug for this episode of AF
* Subject has any known reversible causes of AF such as alcohol intoxication, pulmonary embolism, hyperthyroidism, acute pericarditis or hypoxemia
* Subject has uncorrected electrolyte imbalance
* Subject has clinical evidence of digoxin toxicity
* Subject has a history of clinically significant illness (e.g. neurological, gastrointestinal, renal, hepatic, pulmonary, metabolic, endocrine, hematological, or psychiatric), medical condition or laboratory abnormality within 4 weeks prior to Screening

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2009-10; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Number of Participants who Experience Hypotension, Ventricular Arrhythmias and/or Death | Occurring within the first two hours after start of study treatment
  Hypotension defined as: systolic blood pressure (SBP) <90 mmHg and treated with pressors; SBP <90 mmHg and treated with albumin, dextran or hydroxyethyl starch; or SBP <90 mmHg and seizures. Ventricular arrhythmias defined as: Sustained ventricular tachycardia with a heart rate of >120 beats per minute. Sustained tachycardia defined as lasting >30 seconds; Torsade de Pointes with a duration of >10 seconds; Ventricular fibrillation of any duration.
Number of Participant with Successful Conversion to Sinus rhythm (SR) | Occurring within 90 minutes of first exposure to study treatment
  Successful conversion defined as return to sinus rhythm for at least 1 minute documented by Holter electrocardiogram (ECG) or by two consecutive 12-lead ECGs recorded > 1 minute apart within 90 minutes of first exposure to study treatment

SECONDARY OUTCOMES:
Time from First Exposure to Study Treatment to Conversion of AF to SR | Occurring within 90 minutes after study treatment
Number of Participants who Report No Symptoms | Occurring 90 minutes after first exposure to study treatment
  Participant was considered a success (no symptoms) if they did not have any of the following symptoms at 90 minutes: palpitations, dyspnea, dizziness, chest pain or fatigue

REFERENCES:
- [Derived] Beatch GN, Mangal B. Safety and efficacy of vernakalant for the conversion of atrial fibrillation to sinus rhythm; a phase 3b randomized controlled trial. BMC Cardiovasc Disord. 2016 May 28;16:113. doi: 10.1186/s12872-016-0289-0. PMID 27233239